CLINICAL TRIAL: NCT02534948
Title: Feasibility Study of Mindfulness and Acceptance Based Group Therapy for Females With Social Anxiety
Brief Title: Feasibility Study of Mindfulness and Acceptance Based Group Therapy for Social Anxiety
Acronym: MABT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Zohra Batool, M. Phil Candidate, Bahria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MABT001
Record Dates: First submitted 2015-08-26; First posted 2015-08-28 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Social Anxiety
Keywords: mindfulness; MABT; social anxiety; mindfulness and acceptance; group therapy
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness and acceptance group therapy (Experimental): The intervention group will consist of female participants who will be provided MABT in a group.The intervention will consist of 10 group therapy sessions. Each session will be conducted for 120 minutes.
  Interventions: Behavioral: Mindfulness and acceptance group therapy
- wait list control group (No Intervention): The control group will be the waiting list control group will receive no interventions in the first stage.

INTERVENTIONS:
Behavioral: Mindfulness and acceptance group therapy — The manual group intervention will be provided as per the second edition of Mindfulness and Acceptance-Based Group Therapy for Social Anxiety Disorder: A Treatment Manual developed by Fleming, and Kocovski (2014). The intervention will consist of 10 group therapy sessions. Each session will be conducted in 120 minutes. It includes therapist manual, client handouts, and is written to be used in conjunction with The Mindfulness and Acceptance Workbook for Social Anxiety and Shyness. The treatment manual can be easily adapted for individual therapy clients.
  Arms: Mindfulness and acceptance group therapy

SUMMARY:
Anxiety and depressive disorders are common in all regions of the world. Anxiety disorders are considered as third major psychological issue in Pakistan (Panhwer, 2014). Objective of the present study is to see the feasibility and effectiveness of social anxiety in females with the help of mindfulness and acceptance based therapy. It is hypothesized that women in the intervention group will have significantly reduced anxiety as compared to the women in the control group. A total of 60 females in the age range of 18 to 28 ages will be selected from Institute of professional psychology and private clinics from Karachi city. The participants will be recruited through the administration of Mini-Social Phobia Inventory (SPIN-mini). The participants will be randomly divided in interventions and control group and will receive the intervention of ten sessions of group therapy of MABT plan. Assessment will be conducted at the baseline and at the end of the intervention.

DETAILED DESCRIPTION:
Anxiety and depressive disorders are becoming the major psychological issue in Pakistan due to several circumstances. Social anxiety is one the prominent symbol for psychological disturbance observed in young generation. Since, other therapeutic approaches for social anxiety have not shown significant benefit regarding improvement of symptoms recovery and to avoid relapse of the symptoms, further researches needed to focus on improving post-functioning recovery. The uses of mindfulness and acceptance base group therapy manual for social anxiety has shown significantly reduce symptoms of social anxiety after the therapy in other regions of the world. In this regard the present study will help to enhance the variety of treatment plan and to evaluate the effectiveness of mindfulness in this subject. Therefore, objective of the present study is to see the feasibility and effectiveness of social anxiety in females with the help of mindfulness and acceptance based therapy. In this regard hypothesis is designed as; women in the intervention group will have significantly reduced anxiety as compared to the women in the control group . A total of 60 females in the age range of 18 to 28 ages will be recruited from Institute of professional psychology . The participants will be recruited through the administration of Mini-Social Phobia Inventory (SPIN-mini). Total of 32 participants will be randomly divided in interventions and control group will receive the intervention of ten sessions of group therapy of MABT plan. The manual group intervention will be provided as per the second edition of Mindfulness and Acceptance-Based Group Therapy for Social Anxiety Disorder: A Treatment Manual developed by Fleming, and Kocovski (2014). The intervention will consist of 10 group therapy sessions. Each session will be conducted in 120 minutes. It includes therapist manual, client handouts, and is written to be used in conjunction with The Mindfulness and Acceptance Workbook for Social Anxiety and Shyness. The treatment manual can be easily adapted for individual therapy clients.At the end scores of re-administration of the questionnaire will help to assess the outcomes of the study. Results of this intervention study will be analysed through quantities measures.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who score 6 or above on social phobia inventory.
* Participants who understand Basic English and Urdu language.

Exclusion Criteria:

* History of severe mental illness or organic brain damage i.e. schizophrenia and related disorders; especially in the last few years. Any related medication taken or medication being taken now in this regard.
* Active or recent physical addiction to alcohol or drugs.
* Individuals who were diagnosed with Post-traumatic stress disorder.
* Individuals with severe social anxiety which would make attending very stressful.
* Individuals with already receiving psychological therapy or any other psychiatric treatment.
* Individuals who are involved in persistent self-harm or suicide risk requiring management.

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Mini Social Phobia inventory | three months
  It is a brief screening assessment for generalized social anxiety disorder comprised on 3-item self-rated scale.

CONTACTS AND LOCATIONS:
Overall Officials: Zainab F. Zadeh, Phd, Study Director — Institute of Professional Psychology, Bahria University
Locations (1):
- Institute of Professional Psychology, Bahria University, Karachi, Sindh, Pakistan